CLINICAL TRIAL: NCT00980161
Title: The Predictive Role of Serum Micro RNA-122 to the Clinical Course of Chronic Hepatitis C Patients
Brief Title: Micro RNA-122 and the Clinical Course of Patients With Chronic Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Chen-Hua Liu, National Taiwan University Hospital
Other Study IDs: 200908039R
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Peginterferon; Ribavirin; MicroRNA
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and hepatic micro RNA-122
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Peg-IFN + RBV with SVR: HCV patients receiving peginterferon alfa-2a and ribavirin with sustained virologic response
- Peg-IFN + RBV without SVR: HCV patients receiving peginterferon alfa-2a and ribavirin without sustained virologic response

SUMMARY:
Combination therapy with peginterferon plus ribavirin has become the current standard of care for chronic hepatitis C (CHC) patients, with an overall sustained virologic response (SVR) rate of 54-63%. Based on the ample evidence, a 48-week course of peginterferon plus weight-based ribavirin therapy is widely recommended to treat HCV genotype 1 infection in different parts of the world. Despite the increased SVR rates with the improved medical therapies, about 25-50% and 10-20% of HCV genotype 1 and HCV genotype 2/3 patients may experience relapse after the cessation of therapy with undetectable HCV viremia at the end of treatment. Moreover, combination therapy is costly and may cause various adverse events. Therefore, individualized therapy based on outcome analysis should be adopted to save medical cost as well as to lessen inadequate treatment. Few studies are aimed to evaluate the host responses of micro RNA regulation during interferon-based therapy and its relationships to the overall treatment responses.

Micro RNA (miRNA) is a single-stand RNA composed of 21-23 nucleotides, which may regulate the function of messenger RNA (mRNA). The regulating mechanisms involving micro RNA between the hosts and the HCV virus include (1) auto-regulation of HCV mRNA by HCV miRNA; (2) regulation of host mRNA by HCV miRNA; and (3) regulation of HCV mRNA by host miRNA. MiR-122 is the abundant liver-specific miRNA which is crucial for efficient HCV replication in culture Huh7 cells stably expressing HCV replicons. Recently, an in vivo study for hepatic miR-122 of 42 patients with CHC who received IFN-based therapy showed that patients who did not respond to IFN therapy had markedly decreased pretreatment miR-122 levels. Although miR-122 is abundant in the liver, liver biopsy is still considered an invasive procedure, which prevents its widespread use in routine clinical practice. The miRNA can be detected in the sera and is stable after 24 hours of room temperature store or repeated freezing and de-freezing. The serum miR-122 levels can reflect the severity of liver injuries in a rat acetaminophen toxicity model. Because miR-122 is liver specific and the miRNA is stable in the sera, the investigators aimed to evaluate the role of serum and hepatic miR-122 on the viral kinetics and the treatment responses and in HCV patients receiving peginterferon and ribavirin combination therapy.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection, a leading cause of cirrhosis, hepatocellular carcinoma (HCC) and liver transplantation, affects approximately 170 million individuals worldwide. In Asian-Pacific regions, the prevalence of HCV infection ranges from 0.3-12%, with a geographical variation. Therefore, prevention of HCV transmission and early intervention of HCV infection are urgently needed to reduce or halt the liver-related morbidity and mortality.

Combination therapy with peginterferon plus ribavirin has become the current standard of care for chronic hepatitis C (CHC) patients, with an overall sustained virologic response (SVR) rate of 54-63%. Treatment with weekly peginterferon and weight-based ribavirin for 48 weeks had a significantly higher SVR rate than that for 24 weeks in Caucasian patients with HCV genotype 1 infection (52% to 42%). Based on ample evidence from Western countries, a 48-week course of peginterferon plus weight-based ribavirin therapy is widely recommended to treat HCV genotype 1 infection in different parts of the world. However, recent studies for Asian CHC genotype 1 patients showed favorable treatment response to Caucasian patients with either 24 or 48 weeks of peginterferon plus weight-based ribavirin therapy (50 to 60% for 24 weeks; 75 to 80% for 48 weeks). In contrast, the overall SVR rates were similar across different ethnicity in patients with HCV genotype 2/3 infection.

Despite the increased SVR rates with the improved medical therapies, about 25-50% and 10-20% of HCV genotype 1 and HCV genotype 2/3 patients may experience relapse after the cessation of therapy with undetectable HCV viremia at the end of treatment. Moreover, combination therapy is costly and may cause various adverse events. Therefore, individualized therapy based on outcome analysis should be adopted to save medical cost as well as to lessen inadequate treatment. Currently, HCV viral kinetics is considered to predict treatment response. Patients with rapid virologic response (RVR) are good predictors of SVR; those who fail to achieve RVR but achieve complete or partial early virologic response (cEVR or pEVR) should be put on prolonged therapy; those who fail to achieve EVR should be considered for treatment discontinuation because of low chance for SVR. Various host and viral factors, including race, gender, body weight, baseline viral load, and viral genotype, were considered to predict RVR. However, few studies are aimed to evaluate the host responses of micro RNA regulation during interferon-based therapy and its relationships to the overall treatment responses.

Micro RNA (miRNA) is a single-stand RNA composed of 21-23 nucleotides, which may regulate the function of massager RNA (mRNA). The regulating mechanisms involving micro RNA between the hosts and the HCV virus include (1) auto-regulation of HCV mRNA by HCV miRNA; (2) regulation of host mRNA by HCV miRNA; and (3) regulation of HCV mRNA by host miRNA. MiR-122 is the abundant liver-specific miRNA which is crucial for efficient HCV replication in culture Huh7 cells stably expressing HCV replicons. This observation raised much interest in the role of mir-122 in HCV infection and its potential as a therapeutic target. It was recently reported that the levels of miR-122 and several other miRNAs are regulated by IFN in Huh7 cells and primary mouse hepatocytes and that miRNAs might mediate at least some effects of IFN on HCV RNA replication in vitro. Recently, an in vivo study for hepatic miR-122 of 42 patients with CHC who received IFN-based therapy showed that patients who did not respond to IFN therapy had markedly decreased pretreatment miR-122 levels. Although miR-122 is abundant in the liver, liver biopsy is still considered an invasive procedure, which prevents its widespread use in routine clinical practice. Considering the abundant blood flow through the liver, we speculated that miR-122 can be detected in the sera, and can be used for screening and monitoring the responses by serial blood tests. The miRNA can be detected in the sera and is stable after 24 hours of room temperature store or repeated freezing and de-freezing. In addition, miRNA is resistant to RNase and can be sustained for more than 10 years after adequate freezing. Recent studies have shown the serum miRNA was potentially useful for the detection of cancer and its treatment responses. Furthermore, the serum miR-122 levels can reflect the severity of liver injuries in a rat acetaminophen toxicity model. Because miR-122 is liver specific and the miRNA is stable in the sera, the investigators aimed to evaluate the role of serum and hepatic miR-122 on the viral kinetics and the treatment responses and in HCV patients receiving peginterferon and ribavirin combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve
* Age 18 and older than 18 years old
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum quantitative HCV-RNA (Cobas Taqman v2.0, Roche Diagnostics)
* Serum alanine aminotransferase levels above the upper limit of normal with 6 months of enrollment
* A liver biopsy consistent with the diagnosis of chronic hepatitis C
* Receive 24 or 48 weeks of PEG-IFN alfa plus ribavirin (1,000 mg/day for BW < 75 kg; 1,200 mg/day for BW ≥ 75 kg for HCV genotype 1; 800 mg/day for HCV genotype 2)

Exclusion Criteria:

* Anemia (hemoglobin < 13 gram per deciliter for men and < 12 gram per deciliter for women)
* Neutropenia (neutrophil count <1,500 per cubic milliliter)
* Thrombocytopenia (platelet <90,000 per cubic milliliter)
* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Mixed HCV genotype 1 with other genotype infection
* Chronic alcohol abuse (daily consumption > 20 gram per day)
* Decompensated liver disease (Child-Pugh class B or C)
* Serum creatinine level more than 1.5 times the upper limit of normal
* Autoimmune liver disease
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception
* Without definite viral information during the study period (sustained viral responders or viral relapsers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C receving combination therapy with peginterferon alfa-2a and ribavirin
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Serum micro RNA-122 and sustained virologic response (SVR) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Chair — National Taiwan University Hospital; Jia-Horng Kao, MD, PhD, Study Director — National Taiwan University Hospital; Tung-Hung Su, MD, Principal Investigator — Kimmen Hospital; Cheng-Chao Liang, MD, BS, Principal Investigator — Far Estern Menorial Hospital; Chih-Lin Lin, MD, BS, Principal Investigator — Taipei Municipal Hospital, Ren-Ai Branch; Shih-Jer Hsu, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (5):
- Taiwan (5):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Kinmen Hospital, Kimmen
  - National Taiwan University Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Taipei Municipal Hospital, Ren-Ai Branch, Taipei